CLINICAL TRIAL: NCT02589587
Title: Enteroendocrine Cells in Lean Controls and Healthy Subjects Before and After Sleeve Gastrectomy
Brief Title: Enteroendocrine Cells Before and After Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EEC
Record Dates: First submitted 2015-09-28; First posted 2015-10-28 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleeve gastrectomy (Active Comparator): Morbidly obese patients scheduled for sleeve gastrectomy will be examined by endoscopy before and 3 months after surgery. Biopsies will be taken from stomach and duodenum.
  Interventions: Procedure: sleeve gastrectomy
- no intervention (Other): Lean, healthy controls will undergo endoscopy and biopsies will be taken from stomach and duodenum.
  Interventions: Other: no intervention

INTERVENTIONS:
Procedure: sleeve gastrectomy — Sleeve gastrectomy is an established form of bariatric (weight reducing) surgery, where the greater curvature of the stomach is removed.
  Arms: sleeve gastrectomy
Other: no intervention — lean control group
  Arms: no intervention

SUMMARY:
Morbidly obese patients exhibit impaired secretion of satiation hormones which may contribute to the development of obesity. Bariatric surgery is associated with weight loss and dramatic increase in the secretion of satiation hormones, but the underlying mechanism remains unknown. The investigator's goal is therefore to examine patients before and after sleeve gastrectomy and compare findings to lean controls.

DETAILED DESCRIPTION:
Morbidly obese patients exhibit impaired secretion of satiation hormones cholecystokinin (CCK), glucagon-like peptide 1 (GLP-1) and peptide YY (PYY), which may contribute to the development of obesity. Bariatric surgery is associated with weight loss and dramatic increase in the secretion of satiation hormones, but the underlying mechanism remains unknown. A better understanding of mechanisms involved will assist in development of non-invasive therapeutic strategies. The investigator's goal is therefore to examine patients before and after sleeve gastrectomy and compare findings to lean controls. Gastric and intestinal mucosa will be collected by endoscopy from morbidly obese subjects before and 3 months after sleeve gastrectomy. In Addition, lean controls will be examined. Expression of various gut peptides will be assessed by immunohistochemistry and quantitative polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

Morbidly obese patients scheduled for sleeve gastrectomy

* BMI > 35 kg/m2
* Age: > 18-65 years Lean, healthy controls
* BMI > 18 and < 28kg/m2
* Age: >18-40 years

Exclusion Criteria:

* Bleeding diathesis
* Previous surgery on the gastrointestinal tract (appendectomy acceptable)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quantification of the enteroendocrine cell population | within 3 months after surgery
  Expression of enteroendocrine cell population possessing chromogranin A, ghrelin, CCK, PYY, GLP-1 and GLP-2 by immunohistochemistry and quantitative PCR.

SECONDARY OUTCOMES:
Determination of tissue morphology (crypt depth, villus height) | within 3 months after surgery
  Morphometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided